CLINICAL TRIAL: NCT01614158
Title: Pilot SINN; Assessment of Visual Field (vf)-Related Endpoints in Patients With Non-arteritic Ischemic Optic Neuropathy (N-AION)
Brief Title: Assessment of Visual Field-related Endpoints in Patients With Non-arteritic Ischemic Optic Neuropathy
Acronym: Pilot-SINN
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Ulrich Schiefer, Professor Dr. med. Ulrich Schiefer, University Hospital Tuebingen
Other Study IDs: 73/2009B02
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Non-arteritic Ischemic Optic Neuropathy
Keywords: N-AION; perimetry; visual field loss; Mean Defect; Total Loss Volume; D-BCVA; RAPD; retinal nerve fibre thickness/volume; optic nerve head
MeSH Terms: interventions — Visual Field Tests; Tonometry, Ocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute N-AION (< 7 d): physical, intellectual and linguistic abilities, in order to understand the test requirements
  * willingness to comply with the protocol (4 visits)
  * 45 - 80 years, informed consent
  * acute N-AION (< 7 d)
  * D-BCVA > 0.1 (2/20)
  * RAPD ≥ 0.3 logE steps (neutral density filters)
  Interventions: Device: perimetry; Other: D-BCVA; Other: RAPD; Device: IOP; Device: Spectralis OCT; Other: Fundus photography

INTERVENTIONS:
Device: perimetry — perimetric examination using static stimuli, assessing the entire (80 degree) visual field with a fast thresholding algorithm (GATE) [Schiefer 2008] to know the extent/ magnitude of the visual field defect and its variability within the cohort and over time
  Other Names: Static Perimetry, Octopus 101, thresholding algorithm
Other: D-BCVA — D-BCVA using EDTRS chart
  Other Names: Best Corrected Visual Acuity, EDTRS Chart
Other: RAPD — RAPD using swinging flashlight test
  Other Names: SWIFT-Test
Device: IOP — IOP using applanation tonometer
  Other Names: intraocular pressure
Device: Spectralis OCT — RNFT and RNFV using Spectralis OCT (star scan, ring scan 2,8 mm and volume scan)
  Other Names: RNFT, RNFV, volume scan, star scan, Spectralis OCT
Other: Fundus photography — Optic disk morphology will be documented by fundus photography

SUMMARY:
This present research project intends to collect five quantitative test series:

* perimetric examination using static stimuli, assessing the entire (80 degree) visual field with a fast thresholding algorithm (GATE) [Schiefer 2008] to know the extent/ magnitude of the visual field defect and its variability within the cohort and over time
* D-BCVA, using FrACT [Bach 2007] and EDTRS chart [Ferris 1982]
* RAPD (using swinging flashlight test).
* IOP (using applanation tonometer)
* RNFT and RNFV using Spectralis OCT (star scan, ring scan 2,8 mm, and volume scan) Optic disk morphology will be documented by fundus photography. This assessment of the above-mentioned data is needed in order to allow for estimation of the spontaneous course / fluctuation of the (quantified) functional and morphometric parameters of the N-AION patients during the follow-up period. This is essential for the estimation of the sample size of the subsequently intended SINN study, that is intended to compare different therapeutic strategies in N-AION patients.

ELIGIBILITY:
Inclusion Criteria: - physical, intellectual and linguistic abilities, in order to understand the test requirements

* willingness to comply with the protocol (4 visits)
* 41 - 80 years, informed consent
* acute N-AION (< 7 d)
* D-BCVA > 0.1 (2/20)
* RAPD ≥ 0.3 logE steps (neutral density filters) and:
* spherical ametropia max. ± 8 dpt, cylindrical ametropia max. ± 3 dpt
* isocoria, pupil diameter > 3 mm

Exclusion Criteria:

* diabetic retinopathy and any other orbital, intracranial or optic nerve disease
* history of epilepsy or significant psychiatric disease
* medications known to affect visual field sensitivity
* infections (e.g. keratitis, conjunctivitis, uveitis)
* severe dry eyes
* miotic drug
* amblyopia
* strabismus
* any ocular pathology, in either eye, that may interfere with the ability to obtain visual fields, disc imaging or accurate IOP readings
* cataract with relevant impairment of vision
* keratoconus
* intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening
* history or signs of any visual pathway affection other than N-AION
* history or presence of macular disease and / or macular edema
* ocular trauma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute N-AION (less then 7 days); male and female > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assessment of visual field (VF)-related endpoints in patients with non-arteritic ischemic optic neuropathy (N-AION) | 2 years
  This present research project intends to collect five quantitative test series in order to allow the estimation of the spontaneous course / fluctuation of the (quantified) functional and morphometric parameters of the N-AION patients during the follow-up period. This is essential for the estimation of the sample size of the subsequently intended SINN study, that is intended to compare different therapeutic strategies in N-AION patients

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof., Principal Investigator — Centre for Ophthalmology Institute for Ophthalmic Research University of Tübingen
Locations (1):
- Centre for Ophthalmology Institute for Ophthalmic Research University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Kernstock C, Beisse F, Wiethoff S, Mast A, Krapp E, Grund R, Dietzsch J, Lagreze W, Fischer D, Schiefer U. Assessment of functional and morphometric endpoints in patients with non-arteritic anterior ischemic optic neuropathy (NAION). Graefes Arch Clin Exp Ophthalmol. 2014 Mar;252(3):515-21. doi: 10.1007/s00417-014-2572-z. Epub 2014 Jan 31. PMID 24477537